CLINICAL TRIAL: NCT04308018
Title: Primary Sacroiliac Fusion Versus Fusion to the Sacrum for Degenerative Disease of the Lumbar Spine
Acronym: PSEUDOLUSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20/20
Record Dates: First submitted 2019-11-21; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Degeneration Spine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- S1 (Active Comparator): Caudal end of the instrumentation at S1
  Interventions: Procedure: S1 screws
- S2alar-iliac (Active Comparator): Caudal end of the instrumentation at iliac bone via S2alar-iliac screws
  Interventions: Procedure: S2alar-iliac screws

INTERVENTIONS:
Procedure: S2alar-iliac screws — Caudal end of the instrumentation at iliac bone via S2alar-iliac screws
  Arms: S2alar-iliac
Procedure: S1 screws — Caudal end of the instrumentation at S1
  Arms: S1

SUMMARY:
To prove that the use of additional S2alar-iliac screws for pure lumbar fusions due to degenerative lumbar disease provides superior outcome compared to the standard procedure of fusion to S1.

DETAILED DESCRIPTION:
Patients with symptomatic degenerative spine disease with or without spinal stenosis undergoing lumbosacral fusion to S1. Pedicle screws for posterior Instrumentation and fusion of the lumbar spine plus intervertebral fusion L5/S1 (anterior lumbar inter body fusion (ALIF), transforaminal lumbar inter body fusion (TLIF), or posterior lumbar inter body fusion (PLIF)) with

1. Caudal end of the instrumentation at S1
2. Caudal end of the instrumentation at iliac bone via S2alar-iliac screws

Stratification of both groups by:

* Number of instrumented levels
* Sagittal balance (Roussouly type 1+2 vs. 3+4)

Prospective, randomized, controlled, rater-blinded multicentric interventional study with two parallel groups

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic degenerative spine disease with or without spinal stenosis undergoing lumbosacral fusion to S1
* Lumbar or thoracolumbar Instrumentation
* Planned ventral intervertebral fusion (ALIF, TLIF, PLIF) in L5/S1
* Age ≥ 18 years

Exclusion Criteria:

* Scoliosis >20°
* Chronic steroid usage
* Significant co-morbidity influencing the surgical success:

  * Osteoporosis
  * Rheumatoid arthritis
  * Mental illness/dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Revision rate | 1 year after surgery
  Revisions rates between groups 1 year after surgery

SECONDARY OUTCOMES:
Inter-group Oswestry disability index (ODI) | 3, 6, 12, and 24 months after surgery
  Difference in Oswestry disability index (ODI) between groups 3, 6, 12, and 24 months after surgery
British Medical Research Council (BMRC) scale | 3, 6, 12, and 24 months after surgery
  BMRC scale 3, 6, 12, and 24 months after surgery
Severe adverse events | 3, 6, 12, and 24 months after surgery
  (Severe adverse events) SAE due to instrumentation (new neurological deficit, infection, vascular complications, etc.)
Back pain intensity | 3, 6, 12, and 24 months after surgery
  Back pain intensity at the visual analogue scale (VAS; 0-10; high scores mean a worse outcome) 3, 6, 12, and 24 months after surgery
Health-related quality of life | 3, 6, 12, and 24 months after surgery
  Health-related quality of life evaluated by the "physical component summary (PCS)" of the short-form (SF)-36 3, 6, 12, and 24 months after surgery
Patient satisfaction | 3, 6, 12, and 24 months after surgery
  Patient satisfaction index 3, 6, 12, and 24 months after surgery
Intra-group Oswestry disability index (ODI) | 3, 6, 12, and 24 months after surgery
  Difference in ODI 3, 6, 12, and 24 months after surgery versus preoperatively within the same group
Revision rate II | 24 months after surgery
  Revisions rates between groups 24 months after surgery
Sacroiliac joint syndrome | 3, 6, 12, and 24 months after surgery
  Clinically apparent sacroiliac joint syndrome (Definition: Effective infiltration of local anesthetic) 3, 6, 12, and 24 months after surgery
Gluteal pain | 3, 6, 12, and 24 months after surgery
  Gluteal pain at the visual analogue scale (VAS; 0-10; high scores mean a worse outcome) 3, 6, 12, and 24 months after surgery
Changes in sagittal balance | 1 and 2 years after surgery
  Changes in sagittal balance (C7 plumb line, pelvic tilt, pelvic incidence, sacral slope, and lumbar lordosis) 1 and 2 years after surgery versus preoperatively within the same group
Progressive degeneration of the adjacent segment | 3, 6, 12, and 24 months after surgery
  Radiological proof of progressive degeneration of the adjacent segment
Surgery duration | Surgery
  Surgery duration
Intraoperative blood loss | Intraoperative
  Intraoperative blood loss
Adverse events | 3, 6, 12, and 24 months after surgery
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Krieg, MD, Principal Investigator — Technical University Munich